CLINICAL TRIAL: NCT00683761
Title: A Phase 1/2 Multi-Center, Safety and Efficacy Study Evaluating Intravenously Administered 131I-TM601 in Patients With Progressive and/or Recurrent Malignant Glioma
Brief Title: A Study of 131I-TM601 in Adults With Recurrent Malignant Glioma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TransMolecular (Industry)
Responsible Party: Susan Stewart, Vice President, Regulatory Affairs, TransMolecular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TM601-008
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: Malignant Glioma; Glioblastoma Multiforme; GBM; Astrocytoma; Oligodendroglioma
Keywords: High grade recurrent glioma; Phase 2; Phase 1; Multi-center; Open label; Multiple dose; Brain Cancer; Brain Tumor; GBM; glioma; glioblastoma; astrocytoma; oligodendroglioma; 131I-TM601; TM601
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms | interventions — Chlorotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 131I-TM601

INTERVENTIONS:
Drug: 131I-TM601 — In the first study phase (Dose Escalation), patients will be assigned to treatment to between 2-5 doses of 131I-TM601 treatment at a treatment dose of 1.2 mCi/kg of lean body mass (in scaled dosing, this will amount to 0.024 mg TM601 peptide/kg of lean body mass), once weekly (for between 2-5 weeks, depending upon dose cohort). The maximum amount of administered radioactivity per infusion is 100 mCi.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of 131I-TM601 in the treatment of adult patients with progressive or recurrent malignant gliomas.

DETAILED DESCRIPTION:
This is a multi-center, open label, non-randomized, Phase 1/2 study evaluating the use of multiple intravenous doses of 131I-TM601 in patients with progressive and/or recurrent malignant glioma.

The study will be conducted in two phases. Prior to initiating treatment as part of this study, patients will be administered a single imaging dose of 131I-TM601, IV, to demonstrate tumor uptake. Only patients demonstrating tumor uptake will remain on the study. During the first, Dose Escalation Phase of the study, eligible patients will be assigned in groups of 3-6 (depending upon the treatment response seen at each dose) to dose cohorts of between 2-5 weekly IV doses of 131I-TM601, with escalation to the next highest dose dependent upon demonstrated tolerance in the previous dosing group. Patients enrolled in the second phase will be assigned to a dose determined by the experience in the first phase.

Patients in both study phases will have safety parameters evaluated continuously throughout the study. Clinical response to 131I-TM601 will be assessed in each study patient at 28 days following the final study dose, and then at quarterly intervals scheduled at 3 month intervals following the first study dose, until disease progression.

ELIGIBILITY:
Inclusion Criteria:

Patients must:

1. Have histologically proven malignant glioma (anaplastic astrocytoma, anaplastic oligodendroglioma or glioblastoma multiforme) which is progressive and/or recurrent after external beam radiation therapy (to at least 50 Gy) ± chemotherapy with or without a history of surgical resection. Patients with previous low grade glioma who progressed after radiotherapy ± chemotherapy and are biopsied and found to have a high grade glioma are eligible. Patients with prior therapy that included interstitial brachytherapy, stereotactic radiosurgery, or local radiopharmaceutical injection must have confirmation of true progressive disease rather than radiation necrosis based upon PET or Thallium scanning or pathological documentation of disease.
2. Have bi-dimensional measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 2 planes on post-contrast MRI.

   Note - a CT scan will be acceptable in place of an MRI only in patients who are unable to undergo an MRI.
3. Be ≥18 years of age.
4. Have a baseline Karnofsky Performance Status (KPS) of ≥60%.
5. Have a Mini Mental State Exam score of ≥ 19.
6. Have a life expectancy, based on the Investigator's judgment, of >3 months.
7. On screening ECG, have a QTc interval of <450 ms.
8. If taking steroids, be on a dose that is stable for at least 5 days prior to the Imaging Dose.
9. Have recovered from the toxicity of all previous therapy prior to enrollment. If the patient has undergone recent major surgery, an interval of at least 3 weeks must have elapsed between the surgery and the date of the Imaging Dose.
10. Have adequate organ and marrow function as defined by serum chemistry evaluations (defined in study protocol).
11. Have a negative serum pregnancy test within 14 days of study drug administration, if female and of child bearing potential.
12. Agree to use an effective form of contraception to avoid pregnancy, if fertile (applicable to both male and female patients).
13. Agree to refrain from nursing, if female.
14. Have signed and dated written informed consent.
15. Be able to comply with treatment plan, study procedures and follow-up examinations.

Exclusion Criteria:

Patients may not:

1. Have a serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety. Examples of medical illnesses include, but are not limited to, the following: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
2. Have a prior malignancy with less than 5-year disease free interval, except for adequately treated basal cell or squamous cell carcinoma of the skin, or in situ cancer of the cervix.
3. Have received radiation treatments ≤ 3 months prior to first study drug administration (Imaging Dose).
4. Have received any cytotoxic chemotherapy, whether conventional or investigational, ≤ 4 weeks prior to receiving the first study drug (Imaging Dose) administration in this study (6 weeks for mitomycin-C or nitrosoureas).
5. Have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to 131I-TM601 e.g. iodine or iodine-containing drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-02 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of multiple doses of intravenously (IV) administered 131I-TM601 in adult patients with progressive and/or recurrent malignant glioma with measurable disease. | Safety will be evaluated throughout the treatment and follow-up phase for all study patients; dose escalation decisions will be based on safety experience for each patient at 21 days following the final treament dose.
The therapeutic efficacy of multiple doses of IV-administered 131I-TM601, as assessed by clinical response, time-to-progression, 6 month progression-free survival and overall survival in adult patients with progressive and/or recurrent malignant glioma. | At six months following first treatment dose, and until disease progression.

SECONDARY OUTCOMES:
Radiation absorbed dose to tumor and normal organs from IV administered 131I-TM601 in a subset of study patients. | Assessments timed within 3 days of study doses.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fink, MD, Principal Investigator — Baylor Health Care System; Adam Mamelak, MD, Principal Investigator — Cedars-Sinai Medical Center; Steven Rosenfeld, MD, Principal Investigator — Columbia University; Jan Drappatz, MD, Principal Investigator — Dana-Farber Cancer Institute; Patrick Wen, MD, Principal Investigator — Dana-Farber Cancer Institute; Jeffrey Olson, MD, Principal Investigator — Emory University; Richard Wahl, MD, Principal Investigator — Johns Hopkins University; Heather Jacene, MD, Principal Investigator — Johns Hopkins University; Antonio Omuro, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Edward Pan, MD, Principal Investigator — Moffitt Cancer Center; Sean Grimm, MD, Principal Investigator — Northwestern University; Jeffrey Raizer, MD, Principal Investigator — Northwestern University; Nimish Mobile, MD, Principal Investigator — University of Rochester; Marc Chamberlain, MD, Principal Investigator — University of Washington; Jay-Jiguang Zhu, MD, Principal Investigator — Tufts Medical Center; John Fiveash, MD, Principal Investigator — University of Alabama at Birmingham; David Schiff, MD, Principal Investigator — University of Virginia; Michael Edgeworth, MD, Principal Investigator — Vanderbilt University; Mark Malkin, MD, Principal Investigator — Medical College of Wisconsin; Maciej Mrugala, MD, Principal Investigator — University of Washington; Steven Chmura, MD, Principal Investigator — University of Chicago; Thomas Gribbin, MD, Principal Investigator — St. Mary's Health Care
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - St. Mary's Health Care, Grand Rapids, Michigan
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Background] Mamelak AN, Jacoby DB. Targeted delivery of antitumoral therapy to glioma and other malignancies with synthetic chlorotoxin (TM-601). Expert Opin Drug Deliv. 2007 Mar;4(2):175-86. doi: 10.1517/17425247.4.2.175. PMID 17335414
- [Background] Mamelak AN, Rosenfeld S, Bucholz R, Raubitschek A, Nabors LB, Fiveash JB, Shen S, Khazaeli MB, Colcher D, Liu A, Osman M, Guthrie B, Schade-Bijur S, Hablitz DM, Alvarez VL, Gonda MA. Phase I single-dose study of intracavitary-administered iodine-131-TM-601 in adults with recurrent high-grade glioma. J Clin Oncol. 2006 Aug 1;24(22):3644-50. doi: 10.1200/JCO.2005.05.4569. PMID 16877732
- [Background] Hockaday DC, Shen S, Fiveash J, Raubitschek A, Colcher D, Liu A, Alvarez V, Mamelak AN. Imaging glioma extent with 131I-TM-601. J Nucl Med. 2005 Apr;46(4):580-6. PMID 15809479
- [Background] Lyons SA, O'Neal J, Sontheimer H. Chlorotoxin, a scorpion-derived peptide, specifically binds to gliomas and tumors of neuroectodermal origin. Glia. 2002 Aug;39(2):162-73. doi: 10.1002/glia.10083. PMID 12112367